CLINICAL TRIAL: NCT07145346
Title: Suzetrigine for Acute Pain Control in Patients With Multiple Rib Fractures: A Randomized Controlled Trial
Brief Title: Suzetrigine for Acute Pain Control in Patients With Multiple Rib Fractures
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Jeffry Nahmias, MD, Chief, Division of Trauma, Burns and Surgical Critical Care, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7663
Record Dates: First submitted 2025-08-14; First posted 2025-08-28 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Rib Fractures
Keywords: blunt chest trauma; rib fractures; Suzetrigine; multimodal pain regimen
MeSH Terms: conditions — Rib Fractures

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blinded, placebo-controlled trial
Who Masked: Participant, Care Provider
Masking Description: Patients will be randomized independently by a third party not involved in patient care or data extraction. Researchers and care providers will be blinded to which arm they are in for the duration of the trail.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Suzetrigine arm (Experimental): The intervention arm will receive oral suzetrigine (100 mg loading dose followed by 50 mg every 12 hours).
  Interventions: Drug: Suzetrigine (SUZ)
- Control arm (Placebo Comparator): The control arm will receive placebo capsules matched to suzetrigine for oral administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Suzetrigine (SUZ) — The intervention arm will receive oral suzetrigine (100 mg loading dose followed by 50 mg every 12 hours).
  Arms: Suzetrigine arm
Drug: Placebo — The control arm will receive placebo capsules matched to suzetrigine for oral administration.
  Arms: Control arm

SUMMARY:
Rib fractures cause a significant amount of pain and are associated with an increased risk of lung infections, long hospitalization, and increased cost. Effective pain control is the cornerstone of management to improve lung function and minimize complications. Most often this is done with a multimodal pain routine consisting of: acetaminophen, nonsteroidal anti-inflammatory drugs (NSAIDs), topical lidocaine, muscle relaxants, and opioids. However, suzetrigine is a promising alternative to treat acute pain associated with rib fractures. We think the addition of suzetrigine to a multimodal pain regimen will improve pain and decrease opioid use.

DETAILED DESCRIPTION:
Rib fractures are a common and painful injury associated with increased risk of pneumonia, prolonged hospitalization, and higher healthcare utilization. In a national database review, rib fractures were associated with a 10% mortality rate, with mortality increasing incrementally with each additional rib fractured. Effective analgesia is essential in management of these injuries, as improved pain control optimizes pulmonary mechanics and reduces complications. Current analgesic strategies include multimodal pain regimens consisting of oral and transdermal analgesics or regional anesthetics such as epidural catheters. Historically, opioids have been a major component of analgesia, however they are highly addictive and can lead to respiratory depression and epidurals are invasive procedures with associated risks.

Suzetrigine (Journavx) is a newly United States Food and Drug Administration (FDA)-approved, oral non-opioid analgesic that selectively inhibits the NaV1.8 voltage-gated sodium channel, which is solely expressed in peripheral nociceptive neurons. A systematic review including multiple phase III trials demonstrated suzetrigine's efficacy for pain management in both non-surgical and post-surgical patients. Suzetrigine has also been shown to have comparable analgesia to oral opioids with fewer side effects, such as nausea, vomiting, and need for rescue pain medication.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Blunt trauma patients
* > 3 rib fractures
* Able to tolerate oral intake

Exclusion Criteria:

* < 17 years old
* Pregnant
* Prisoners
* History of adverse reaction to suzetrigine
* Current strong CYP3A inhibitor medication use

  o Strong Inhibitors: clarithromycin, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, atazanavir, darunavir, indinavir, lopinavir, telithromycin
* Current strong or moderate CYP3A inducer

  * Strong Inducers: apalutamide, carbamazepine, encorafenib, enzalutamide, fosphenytoin, lumacaftor and ivacaftor, mitotane, phenytoin, rifampin
  * Moderate Inducers: bexarotene (Systemic), bosentan, cenobamate, dabrafenib, dipyrone, efavirenz, elagolix, estradiol, and norethindrone, eslicarbazepine, etravirine, fexinidazole, lorlatinib, mitapivat, modafinil, nafcillin, pacritinib, pexidartinib, phenobarbital, primidone, repotrectinib, rifabutin, rifapentine, sotorasib, St John's Wort
* Cirrhosis
* GCS < 14
* Rhabdomyolysis (CPK > 5,000 U/L)
* Chronic opioid use (>30mg OME/day)
* Known or suspected active infection with human immunodeficiency virus or hepatitis B or C viruses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Pain | Through study completion of index hospitalization (up to 2 years)
  Pain will be measured on a numerical pain scale from 0 (no pain) to 10 (most pain). Higher pain scores equate to worse outcomes.
Use of morphine and morphine equivalents | Through study completion of index hospitalization (up to 2 years)
  Oral morphine equivalents (OME) - A study team member will do a chart review and collect morphine used by the patients.

SECONDARY OUTCOMES:
Epidural Administration | Through study completion of index hospitalization (up to 2 years)
  Epidural use - patients that fail pain management will be offered an epidural
Time in the Hospital | Through study completion of index hospitalization (up to 2 years)
  ICU length of stay - number of days in the ICU Hospital length of stay - number of days admitted to the acute care hospital
Respiratory Complications | Through study completion of index hospitalization (up to 2 years)
  Respiratory complications - include events such as unplanned intubation, pneumonia, pneumothorax and incentive spirometry
Mortality | Through study completion of index hospitalization (up to 2 years)
  Mortality - in-hospital mortality rate and 30-day mortality

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Irvine, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galvagno SM Jr, Smith CE, Varon AJ, Hasenboehler EA, Sultan S, Shaefer G, To KB, Fox AD, Alley DE, Ditillo M, Joseph BA, Robinson BR, Haut ER. Pain management for blunt thoracic trauma: A joint practice management guideline from the Eastern Association for the Surgery of Trauma and Trauma Anesthesiology Society. J Trauma Acute Care Surg. 2016 Nov;81(5):936-951. doi: 10.1097/TA.0000000000001209. PMID 27533913
- [Background] Stawicki SP, Grossman MD, Hoey BA, Miller DL, Reed JF 3rd. Rib fractures in the elderly: a marker of injury severity. J Am Geriatr Soc. 2004 May;52(5):805-8. doi: 10.1111/j.1532-5415.2004.52223.x. PMID 15086666
- [Background] Bulger EM, Arneson MA, Mock CN, Jurkovich GJ. Rib fractures in the elderly. J Trauma. 2000 Jun;48(6):1040-6; discussion 1046-7. doi: 10.1097/00005373-200006000-00007. PMID 10866248
- [Background] Carver TW, Kugler NW, Juul J, Peppard WJ, Drescher KM, Somberg LB, Szabo A, Yin Z, Paul JS. Ketamine infusion for pain control in adult patients with multiple rib fractures: Results of a randomized control trial. J Trauma Acute Care Surg. 2019 Feb;86(2):181-188. doi: 10.1097/TA.0000000000002103. PMID 30376537
- [Background] Schnabel A, Meyer-Friessem CH, Reichl SU, Zahn PK, Pogatzki-Zahn EM. Is intraoperative dexmedetomidine a new option for postoperative pain treatment? A meta-analysis of randomized controlled trials. Pain. 2013 Jul;154(7):1140-9. doi: 10.1016/j.pain.2013.03.029. Epub 2013 Mar 27. PMID 23706726
- [Background] Peng K, Zhang J, Meng XW, Liu HY, Ji FH. Optimization of Postoperative Intravenous Patient-Controlled Analgesia with Opioid-Dexmedetomidine Combinations: An Updated Meta-Analysis with Trial Sequential Analysis of Randomized Controlled Trials. Pain Physician. 2017 Nov;20(7):569-596. PMID 29149140
- [Background] Zhang X, Wang D, Shi M, Luo Y. Efficacy and Safety of Dexmedetomidine as an Adjuvant in Epidural Analgesia and Anesthesia: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Clin Drug Investig. 2017 Apr;37(4):343-354. doi: 10.1007/s40261-016-0477-9. PMID 27812971
- [Background] Gerlach AT, Murphy CV, Dasta JF. An updated focused review of dexmedetomidine in adults. Ann Pharmacother. 2009 Dec;43(12):2064-74. doi: 10.1345/aph.1M310. PMID 19934395
- [Background] Flagel BT, Luchette FA, Reed RL, Esposito TJ, Davis KA, Santaniello JM, Gamelli RL. Half-a-dozen ribs: the breakpoint for mortality. Surgery. 2005 Oct;138(4):717-23; discussion 723-5. doi: 10.1016/j.surg.2005.07.022. PMID 16269301